CLINICAL TRIAL: NCT05039567
Title: The Effect of an Optimal Heart Team Implementation Protocol on the Stability of Decision-making for Complex Coronary Artery Disease-a Randomized Controlled Trial
Brief Title: Effect of an Optimal Heart Team Protocol on Decision-making Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1303-2
Record Dates: First submitted 2021-08-26; First posted 2021-09-09 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
Keywords: Heart Team protocol; Coronary Artery Disease; decision-making agreement
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- optimal heart team group (Experimental): Heart teams in this group will be established according to the optimal heart team protocol. Each team consists of two interventional cardiologists and two cardiac surgeons. Team members will be trained systematically before the heart team meeting.
  Interventions: Behavioral: optimal heart team protocol
- conventional heart team group (No Intervention): Heart teams in this group will be established according to the basic elements recommended by guidelines. Each team consists of an interventional cardiologist, a cardiac surgeon, and a non-interventional cardiologist. No team training will be held before the heart team meeting.

INTERVENTIONS:
Behavioral: optimal heart team protocol — Heart teams in the experimental group will be established and trained based on the optimal heart team implementation protocol. The protocol included instructions on specialist selection, specialist training, team composition, team training and formal implementation precess.
  Arms: optimal heart team group

SUMMARY:
This study is aimed to evaluate the effect of the optimal heart team implementation protocol on the stability of decision-making for patients with complex coronary artery disease.

DETAILED DESCRIPTION:
Current guidelines recommend a heart team in the decision making for patients with complex coronary artery disease (CAD). Previous study reported that the agreement between heart teams for revascularization decision-making in complex CAD patients was moderate. Potential factors associated with decision discrepancies were summarized in several aspects and a detailed heart team implementation protocol was generated and further validation is needed. This study is designed to evaluate the effect of the optimal heart team implementation protocol on the stability of decision-making for patients with complex coronary artery disease.

ELIGIBILITY:
Eligibility Criteria for patients:

Inclusion Criteria:

Patients with stable CAD according to the National Cardiovascular Data Registry (NCDR) CathPCI criteria (stable angina, no or silent myocardial ischemia) and angiographically confirmed 3-vessel disease or left main disease.

Exclusion Criteria:

1. prior percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG);
2. cardiac troponin I (CTnI) greater than the local laboratory upper limit of normal or recent myocardial infarction with CTnI levels still elevated;
3. concomitant severe valvular disease, macrovascular disease, or huge ventricular aneurysm requiring surgery;
4. concomitant atrial fibrillation or severe arrhythmia

Eligibility Criteria for specialists:

Inclusion Criteria for interventional cardiologists:

1. Annual PCI volume ≥200
2. Annual left main PCI volume ≥25
3. Capable of chronic total occlusion(CTO) PCI
4. Clinical researcher experience in coronary revascularization
5. Proficient in clinical guidelines

Inclusion Criteria for cardiac surgeons:

1. CABG total volume ≥200
2. Proficient in both on-pump and off-pump CABG
3. Clinical researcher experience in coronary revascularization
4. Proficient in clinical guidelines

Inclusion Criteria for non-interventional cardiologists:

1) Proficient in clinical guidelines

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Overall percent agreement | through study completion, an average of 1 year
  The proportion of patients who received unanimous decision recommendations from the heart team

SECONDARY OUTCOMES:
Kappa value of heart team decision-making | through study completion, an average of 1 year
  Fliess's (more than 2 raters) and Cohen's (2 raters) kappa coefficients to evaluate inter-team, inter-specialist, and inter-round agreement for treatment decisions.
Inappropriate decision rate | through study completion, an average of 1 year
  According to the American College of Cardiology/American Association for Thoracic Surgery/American Heart Association 2017 Appropriate Use Criteria for coronary revascularization, the inappropriate decision rate od decision-making
Compliance rate in real-world treatment | through study completion, an average of 1 year
  Compliance is defined as the patient's actual treatment meeting the recommendations of either heart team
Reproducibility of decision-making | At 1-month after first phase of heart team meeting
  All cases will be discussed by the same heart team to evaluate the intra-team consistency in decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Zheng, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- National Clinical Research Center for Cardiovascular Diseases, State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma H, Lin S, Li X, Wang Y, Xu B, Zheng Z. Effect of a standardised heart team protocol versus a guideline-based protocol on revascularisation decision stability in stable complex coronary artery disease: rationale and design of a randomised trial of cardiology specialists using historic cases. BMJ Open. 2022 Dec 1;12(12):e064761. doi: 10.1136/bmjopen-2022-064761. PMID 36456006